CLINICAL TRIAL: NCT05933915
Title: The Effect of Laughter Yoga on the Secondary Traumatic Stress Level and Psychological Well-Being of Midwives
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Assoc. Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBU-AYDINKARTAL002
Record Dates: First submitted 2023-06-24; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Laughter Yoga
Keywords: laugh; yoga; secondary trauma; psychological well-being
MeSH Terms: conditions — Laughter; Compassion Fatigue; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Single blind randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Laughter yoga group) (n:40) (Experimental): Laughter yoga will be practiced to midwives in the intervention group.
  Interventions: Other: group-based laughter yoga
- Control Group (n:40) (No Intervention): The control group will not be subjected to any application.

INTERVENTIONS:
Other: group-based laughter yoga — Midwives in the intervention group of the research will apply 8 sessions of laughter yoga, 2 sessions a week. Laughter yoga will be practiced by researchers with leadership certification. Each session will take an average of 45 minutes. Laughter Yoga sessions will be held on the web through the "Zoom" program. Each session will consist of groups of 8 people.
  Arms: Intervention Group (Laughter yoga group) (n:40)

SUMMARY:
Aim: The aim of this study is to determine the effect of laughter yoga, which includes various relaxing practices, on secondary trauma levels and psychological well-being of midwives. The study was planned as a randomized controlled experimental study. This RCT will be administered following the CONSORT 2010 guidelines.

Material and Methods: Considering the case losses in the study, it was planned to create a total of 80 midwives, 40 in the intervention group and 40 in the control group. Laughter yoga will be practiced in the intervention group. No intervention will be made on the control group. Data were collected by using the Personal Information Form, Secondary Traumatic Stress Scale, Psychological Well-Being Scale.

DETAILED DESCRIPTION:
Physiologically, laughter increases blood oxygen saturation, beta endorphin levels increase; It is stated that it has psychological effects such as reducing anxiety, stress, depression and facilitating social communication. Laughter yoga is a non-pharmacological therapy. Laughter yoga is also used to improve general health, reduce mental symptoms, and improve quality of life. Midwives will be randomly assigned to the intervention and control groups, and computer-assisted randomization, one of the fixed probability randomization methods, will be used (https://www.randomizer.org/#randomize). The study will be conducted single-blind. The researcher who will do the laughter yoga and the researcher who will apply the evaluation questionnaires will be different. The researcher who will make the analysis and evaluation will be blind to the groups of midwives.

Midwives in the intervention group of the research will apply 8 sessions of laughter yoga, 2 sessions a week. Laughter yoga will be practiced by researchers with leadership certification. Each session will take an average of 45 minutes. Laughter Yoga sessions will be held on the web through the "Zoom" program. Each session will consist of groups of 8 people. Before starting the laughter yoga, 5 separate WhatsApp groups consisting of 8 people will be established to provide faster and easier communication with the midwives in the intervention group, and communication will be provided by informing and communicating about the sessions. Before starting the application, the "Zoom" program will be downloaded to the phones or computers of the midwives in the intervention group. "Secondary Traumatic Stress Scale" and "Psychological Well-Being Scale" will be applied to midwives before and 4-6 weeks after the application.

Control Group: No intervention will be applied to the control group midwives, and the Secondary Traumatic Stress Scale" and "Psychological Well-Being Scale" will be applied again when they are included in the study and 4-6 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Being a midwifery graduate and working actively in the field
* Volunteering to participate in the research

Exclusion Criteria:

* Any psychiatric diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | Before application
  In this form, which was created by the researchers based on the literature, the participants' age, the high school they graduated from, their willingness to choose the profession, their feeling of belonging to the profession, the unit they work in, their working status in crisis situations, etc. questions are included.
Psychological Well-Being Scale | Before application
  The scale was developed to measure current socio-psychological well-being. Scores that can be obtained from the scale range from 8 (if strongly disagree with all items) to 56 (if strongly agree with all items). It is concluded that individuals with high scores have high psychological resources.
Secondary Traumatic Stress Scale | Before application
  The scale consists of 17 items and is scored with a 5-point Likert-type rating (1=Never, 5=Very often). The scale has three sub-dimensions: emotional violation, avoidance and arousal. Items numbered 2,3,6,10,13 evaluate emotional violation sub-dimension; items numbered 1,5,7,9,12,14,17 evaluate avoidance sub-dimension; items numbered 4,8,11,15,16 evaluate arousal sub-dimension. The score that can be obtained from the scale is between 17 and 85 and the increase in the score indicates a high level of affectivity.

SECONDARY OUTCOMES:
Secondary Traumatic Stress Scale | 4-6 weeks after application
  The scale consists of 17 items and is scored with a 5-point Likert-type rating (1=Never, 5=Very often). The scale has three sub-dimensions: emotional violation, avoidance and arousal. Items numbered 2,3,6,10,13 evaluate emotional violation sub-dimension; items numbered 1,5,7,9,12,14,17 evaluate avoidance sub-dimension; items numbered 4,8,11,15,16 evaluate arousal sub-dimension. The score that can be obtained from the scale is between 17 and 85 and the increase in the score indicates a high level of affectivity.
Psychological Well-Being Scale | 4-6 weeks after application
  The scale was developed to measure current socio-psychological well-being. Scores that can be obtained from the scale range from 8 (if strongly disagree with all items) to 56 (if strongly agree with all items). It is concluded that individuals with high scores have high psychological resources.

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Aydın Kartal Assoc. Prof. Dr., Principal Investigator — Saglik Bilimleri Universitesi; Aleyna Bulut Research Assistant, Study Chair — Saglik Bilimleri Universitesi; Sema Aker Research Assistant, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No